CLINICAL TRIAL: NCT02369029
Title: An Open-label, Non-randomized, Multicenter Phase I Dose Escalation Study to Characterize Safety, Tolerability, Pharmacokinetics and Maximum Tolerated Dose of BAY 1238097 in Subjects With Advanced Malignancies
Brief Title: BAY1238097, First in Man
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17437; 2014-003131-19 (EudraCT Number)
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms
Keywords: Phase I; Dose escalation; NUT-midline carcinoma; Acute Leucemia; Lymphoma; Melanoma; Myeloma; HCC; NSCLC
MeSH Terms: conditions — Neoplasms; Lymphoma; Melanoma; Neoplasms, Plasma Cell | interventions — BAY 1238097

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): To determine maximum tolerated dose (MTD) of BAY 1238097
  Interventions: Drug: BAY 1238097

INTERVENTIONS:
Drug: BAY 1238097 — Oral administration twice weekly. Starting dose will be 10 mg per week and dose will be escalated dependent on any dose limiting toxicities.

SUMMARY:
This is the first study where BAY1238097 is given to humans. Impact of the study is to evaluate if patients with advanced cancer show clinical benefit under the treatment with BET(Bromodomain and extraterminal domain family ) inhibitor.Patients with solid tumors (all comers) and lymphoma will receive the study drug treatment in an escalation scheme (no placebo group) to determine the safety, tolerability and maximum tolerated dose (MTD) of BAY1238097. the relative bioavailability of Liquid Service Formulation and tablets will be determined

After MTD is defined, patients with solid tumors (all comer, hepato cellular carcinoma, lung cancer, NUT(nuclear protein in testis)-midline carcinoma), melanoma and lymphoma will be enrolled A separate escalation scheme will be applied to patients with leucemias, and at the maximal tolerated dose, patients with AML amd multiple myeloma will be enrolled.

the study will also assess the pharmacokinetics, biomarker status, pharmacodynamic parameters of BAY1238097 and tumor response to the treatment.

BAY1238097 will be given twice weekly as oral application. Treatment will be stopped if the tumor continues to grow, if side effects occur, wich the patient cannot tolerate or if the patient decides to withdraw from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, histologically or cytologically confirmed tumor, refractory to any standard treatment, with no standard therapy available, in whom standard therapy is not a therapeutic option or the subject actively refuses use of chemotherapy which would be regarded standard and/or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Adequate liver and renal functions as assessed by the following laboratory requirements to be conducted within 7 days prior to starting study treatment:
* Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN for subjects with hepatic involvement with tumor)
* Amylase and lipase ≤ 2.5 x ULN (≤ 5 x ULN for subjects with pancreas involvement with tumor)
* Prothrombin time (PT-INR)/ partial thromboplastin time (PTT) ≤ 1.5 x ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement that is pre dose as defined by the local standard of care
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min per 1.73 m2 according to the Modification of Diet in Renal Disease Study Group (MDRD) formula (see Section 14.6)
* Adequate cardiac function (left ventricular ejection fraction [LVEF] ≥50% measured by echocardiography or multi-gated acquisition [MUGA] scan)

Exclusion Criteria:

* History of cardiac disease including congestive heart failure New York Heart Association (NYHA) Class >II (Section 14.7), unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months) or myocardial infarction within the past 6 months and cardiac arrhythmias requiring anti-arrhythmic therapy except for beta-blockers and digoxin; evidence for uncontrolled coronary artery disease (eg angina pectoris, myocardial infarction within 6 months prior to study entry, major regional wall motion abnormalities upon baseline echocardiography)
* Moderate and severe hepatic impairment, ie Child-Pugh B or C
* Restrictive lung diseases due to parenchymal damage (eg idiopathic lung fibrosis) or pleural adhesions. Patients with lung resection, scoliosis or thorax malformations can be included provided adequate spirometry testing during screening (eg FEV-Forced expiratory volume 1 ≥ 70%; age, sex and height adapted vital capacity)
* Evidence or history of bleeding diathesis. Any hemorrhage/bleeding event ≥ CTCAE (Common terminology criteria for adverse events) Grade 3 within 4 weeks of first dose of study drug
* Human immunodeficiency virus (HIV) infection
* Chronic or active hepatitis B or C (patients positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA; patients positive for HCVAb will be eligible if negative for HCV-RNA)
* History of other malignancy which could affect compliance with the protocol or interpretation of results. Patients with a history of curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix or breast are allowed. Patients with a malignancy that has been treated with curative intent will also be allowed if the malignancy has been in complete remission without treatment for at least 1 year prior to Cycle 1 Day 1 of study treatment. A recent history of myelodysplastic syndrome in patients with secondary leukemia is allowed
* Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
* Any condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the study
* Anticancer chemotherapy or immunotherapy during the study or within less than 3 half-lives for anticancer chemotherapy or 6 weeks for antibody therapies (2 weeks for leukemia patients) prior to start of study drug.
* Use of any strong CYP3A4 inhibitor such as ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir, or saquinavir (see Table 6 6) 14 days before the first dose of study drug or during the study
* Use of any strong CYP3A4 inducer such as rifampin, St John's Wort, or other herbal preparations that contain any strong CYP3A4 inducer (see Table 6 6) 14 days before the first dose of study drug or during the study
* Clinically relevant findings in the ECG such as a second-degree or third-degree atrioventricular (AV) block (subjects with AV block and pacemaker in place for >1 year and checked by a cardiologist within ≤6 months before the first dose of study drug will not be excluded), prolongation of the QRS complex over 120 msec or of the QTc interval (Fridericia, QTcF) over 470 msec (subjects with a pacemaker and QRS interval over 120 msec or QTc inverval over 470 msec may be enrolled on a case-by-case basis, following a discussion between the investigator and the sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
incidence of DLT(dose-limiting toxicities) | Cycle 1(the first 21 days )

SECONDARY OUTCOMES:
Tumor response evaluation based on the response criteria as applicable | up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Houston, Texas, United States
- HUS, Finland
- Villejuif, France
- Heidelberg, Baden-Wurttemberg, Germany
- Bellinzona, Switzerland
- Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Postel-Vinay S, Herbschleb K, Massard C, Woodcock V, Soria JC, Walter AO, Ewerton F, Poelman M, Benson N, Ocker M, Wilkinson G, Middleton M. First-in-human phase I study of the bromodomain and extraterminal motif inhibitor BAY 1238097: emerging pharmacokinetic/pharmacodynamic relationship and early termination due to unexpected toxicity. Eur J Cancer. 2019 Mar;109:103-110. doi: 10.1016/j.ejca.2018.12.020. Epub 2019 Jan 31. PMID 30711772